CLINICAL TRIAL: NCT01527123
Title: A Study to Evaluate the Pharmacokinetics of Benzoic Acid and Hippuric Acid After Topical Administration of GSK2585823 in Japanese Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 115959
Record Dates: First submitted 2012-01-26; First posted 2012-02-06 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Acne Vulgaris
Keywords: GSK2585823, benzoic acid, hippuric acid, acne vulgaris, pharmacokinetics
MeSH Terms: conditions — Acne Vulgaris

ARMS (1):
- GSK2585823 (Experimental): External Preparation
  Interventions: Drug: GSK2585823

INTERVENTIONS:
Drug: GSK2585823 — CLDM1%/BPO3%

SUMMARY:
This is a Phase 1, single-center, open-label study to evaluate the pharmacokinetics of the BPO metabolites benzoic acid and hippuric acid with 7-day repeat application of GSK2585823 in subjects with acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female subjects between 20 and 45 years of age inclusive at the time of signing the informed consent. Rationale: It is considered as adult and the qualifying maximum age expected of subjects with acne vulgaris with good health.
* Diagnosis of acne vulgaris by a dermatologist. Other than acne vulgaris subject must be in good general condition as determined by a investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. Rationale: It is considered as adult and the qualifying maximum age expected of subjects with acne vulgaris with good health.
* Subjects must have, on the face at screening (physical examination of dermatologist): A minimum of 17 but not more than 60 inflammatory acne lesions (papules / pustules), including nasal lesions; and a minimum of 20 but not more than 150 non-inflammatory acne lesions (open / closed comedones), including nasal lesions. It is set to evaluate acne patients in the same degree of severity of Japanese Phase 3 study.
* A female subject is eligible to participate if she is of: Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up examination. Rationale: It is considered as adult and the qualifying maximum age expected of subjects with acne vulgaris with good health.
* Body weight greater than and equal to 50 kg and body mass index (BMI) within the range greater than and equal to18.5 to less than 29.0 kg/m2 at screening Rationale: It is considered as adult and the qualifying maximum age expected of subjects with acne vulgaris with good health.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. Rationale: It is included from an ethical viewpoint according to GCP.
* Single QTcB less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block. Rationale: It is considered as adult and the qualifying maximum age expected of subjects with acne vulgaris with good health.
* AST, ALT, alkaline phosphatase and total bilirubin les than and equal to ULN at screening. Rationale: It is considered as adult and the qualifying maximum age expected of subjects with acne vulgaris with good health.

Exclusion criteria:

* Have a history or presence of regional enteritis, inflammatory bowel disease (e.g., ulcerative colitis, pseudomembranous colitis, chronic diarrhea, antibiotic-associated colitis or bloody diarrhea) or similar symptoms. Rationale: It is considered necessary to secure subject's safety.
* Pregnant females as determined by positive urine hCG test at screening or lactating females. Rationale: It is considered necessary to secure subject's safety.
* Used any of the following agents on the face within the previous 2 weeks: Topical antibiotics (or systemic antibiotics); Topical anti-acne medications (e.g., BPO, azelaic acid, resorcinol, salicylates); Abradants, facials, or peels containing glycolic or other acids; Masks, washes or soaps containing BPO, sulfacetamide sodium, or salicylic acid; Non-mild facial cleansers (e.g., facial scrub, cleansers containing agents with anti-inflammatory action); Moisturizers that contain retinol, salicylic acid, or α- or β-hydroxy acids; Astringents and toner (Subjects are allowed to enroll in this study, if the subject has been on treatment for more than 2 consecutive weeks prior to start of investigational product use); Topical corticosteroids (Use of inhaled, intra-articular, or intra-lesional steroids other than for facial acne is acceptable); Facial procedure (such as chemical or laser peel, microdermabration, blue light treatment, etc.); Topical retinoids on the face Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Used systemic retinoids within the previous 6 months. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Received treatment with estrogens, androgens, or anti-androgenic agents within the previous 12 weeks (Subjects who have been treated with the above agents for more than 12 consecutive weeks prior to start of investigational product are allowed to enrol as long as they do not expect to change dose, drug, or discontinue use during the study). Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Used any medication that in the opinion of the investigator may affect this clinical study or evaluation of the study. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Have a known hypersensitivity or have had previous allergic reaction to any of the components of the investigational product. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Used any investigational therapy within the previous 4 months, or plan to participate in another clinical study at the same time. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* A positive test for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody at screening. Rationale: To secure the site staffs' safety.
* A positive drug screen at screening. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Participated in Japanese clinical studies planned by GlaxoSmithKline K.K. in the development of investigational products for acne vulgaris. Rationale: To be incompatible with stopping criteria.
* Are currently abusing drugs or alcohol. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study and to avoid the double-count of subjects.
* Have a significant medical history of being immunocompromised. Rationale: It is considered necessary to secure subject's safety and to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* People as follows and the family members; Employees of GlaxoSmithKline, contract research organization (CRO) or site management organization (SMO); Investigators (or subinvestigators). Rationale: : It is considered necessary to secure subject's safety.
* The subject has donated a unit of blood ">400 mL" within the previous 4 months or ">200 mL" within the previous 1 month. Rationale: It is considered necessary to secure subject's safety. It is included from an ethical viewpoint.
* Painters or subjects working at the coating industry including automobile mechanic. Rationale: : It is considered necessary to secure subject's safety.
* Unwillingness or inability to follow the procedures outlined in the protocol. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study and to avoid the subject potentially has high level of blood concentration of benzoic acid.
* Subject is mentally or legally incapacitated. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.
* Have other conditions that would put the subject at unacceptable risk for participation in the study. Rationale: It is considered necessary to appropriately assess the safety and pharmacokinetics of GSK2585823 in the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of plasma benzoic acid and hippuric acid pharmacokinetics between pre-application and post-application (7-days repeat) of GSK2585823 | Participants will be followed up to 7 days after the last application, an expected average of 15 days
  Blood PK sampling time frame: 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9,12hours post-dose (Day 1 and Day 8). Parameters: Maximum observed concentration(Cmax),Time of occurrence of Cmax (tmax), Area under the concentration-time curve from time zero (pre-dose) extrapolated to last time (AUC0-last), Area under the concentration-time curve from time zero (pre-dose) to 12 hours of quantifiable concentration within a subject across all treatments (AUC0-12) and Terminal phase half-life (t1/2,) for both benzoic acid and hippuric acid, after multiple application of GSK2585823, if calculable

SECONDARY OUTCOMES:
Comparison of urine benzoic acid and hippuric acid | Participants will be followed up to 7 days after the last application, an expected average of 15 days
  Urine PK sampling time frame:0-4, 4-8, 8-12 hours post-dose (Day 1 and Day 8). Parameters: Renal clearance (CLr), amount of elimination (Ae) and fraction of elimination (fe), if calculable.
change from baseline in vital signs, ECGs, clinical laboratory tests | Day -1 - Day 15
  Vital signs, ECGs, clinical laboratory tests
Collection of adverse events | Participants will be followed up to 7 days after the last application, an expected average of 15 days
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115959 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115959?search=study&search_terms=115959#rs
- Available data/document: Informed Consent Form: 115959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115959 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register